CLINICAL TRIAL: NCT01873066
Title: An Open-label, Single-centre, Randomised, Two-period Crossover Study to Assess the Efficacy, Safety and Utility of Automated Closed-loop Glucose Control, Day and Night Over 7 Days (Phase 1) and 21 Days (Phase 2) in Comparison With Continuous Subcutaneous Insulin Infusion Combined With Continuous Glucose Monitoring in the Home Setting in Children and Adolescents T1D
Brief Title: Closing the Loop 24/7 in Adolescents With Type 1 Diabetes
Acronym: DAN04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Director of Research, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAN04
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases
Keywords: Type 1 diabetes; Closed-loop glucose control; Artificial Pancreas; Continuous subcutaneous insulin infusion; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed-loop insulin delivery (Experimental): Glucose level is controlled by the automated closed-loop glucose control system. After initial training with the closed-loop system devices, subjects will use the closed-loop system day and night at home for a total duration of 7 days (phase 1) and 21 days (phase 2).
  Interventions: Device: Closed-loop system; Device: real-time CGM
- real-time CGM alone (Active Comparator): Glucose level will be controlled by usual insulin pump therapy in conjunction with real time continuous glucose monitoring (CGM) during the day and night over 7 days (phase 1) and 21 days (phase 2).
  Interventions: Device: real-time CGM

INTERVENTIONS:
Device: Closed-loop system — The closed-loop system is purpose-built and comprises a hand-held computer containing a model predictive control (MPC) based glucose control algorithm and communicating with the CGM device and the insulin pump.
  Arms: Closed-loop insulin delivery
Device: real-time CGM — Subject's glucose level is controlled by usual insulin pump therapy in conjunction with real time continuous glucose monitoring (CGM)

SUMMARY:
Type 1 diabetes (T1D) is one of the most common chronic childhood diseases requiring lifelong insulin therapy. Children and adolescents with T1D need regular insulin injections or the continuous insulin delivery using an insulin pump in order to keep blood glucose levels normal. We know that keeping blood sugars in the normal range will help prevent long-term diabetes-related complications involving the eyes, kidneys and heart. However, achieving treatment goals can be very difficult particularly due to the risk of low glucose levels (hypoglycaemia). One solution is to use a system where the amount of insulin injected closely matches the blood sugar levels on a continuous basis. This can be achieved by what is known as a "closed-loop system" where a small glucose sensor placed under the skin communicates with a computer containing an algorithm that drives a subcutaneous insulin pump. We have been testing such a system in Cambridge over the last five years in children and have found that this system is effective, and superior to usual insulin pump therapy, at maintaining tight glucose control. More recently the system has been tested overnight, in the home setting, for three weeks in adolescents during a pilot single-centre study.

The next step is to evaluate use of the closed loop system day and night over a period of 7 days (phase 1) and 21 days (phase 2) in adolescents with type 1 diabetes. In the present study we are planning to study 24 (12 phase 1 ans 12 phase 2) young people aged 10-18 years on insulin pump therapy. This study will involve two 7 (phase 1) and 21 (phase 2) day home study periods, during which glucose levels will be controlled either by an automated closed-loop system or by subjects usual insulin pump therapy combined with continuous glucose monitoring alone in random order. Prior to the closed-loop study period, there will be a training period in the clinical research facility, which will allow participants to familiarise themselves with the closed-loop system before going home.

We aim to to determine the effect of the closed-loop computer algorithm in keeping glucose levels between 3.9 and 10.0 mmol/L during the daytime and overnight.

DETAILED DESCRIPTION:
The main objective of this study is to determine the efficacy, safety and utility of automated closed-loop glucose control in the home setting over a short term period, including the daytime and during the activities of normal daily living. This study builds on previous and on-going studies of closed-loop systems that have been performed in Cambridge in children and adolescents with type 1 diabetes in the clinical research facility and in the home setting. The data and experienced gained from this study will be utilised in planning future home studies.

This is an open-label, single-centre, randomised, crossover study, involving two, 7 day (phase 1) and 21 day (phase 2) home study periods during which glucose levels will be controlled either by an automated closed-loop system or by subjects' usual insulin pump therapy combined with continuous glucose monitoring in random order. A total of up to 30 children and adolescents aged 10 to 18 years with T1D on insulin pump therapy will be recruited through diabetes clinics, to allow for 12 completed subjects available for assessment in each study phase.

Subjects will receive appropriate training by the research team on the safe use of the closed-loop insulin delivery system. During the training visit in a clinical research centre, subjects will be encouraged to mimic their usual daily activities and will be allowed to walk inside hospital premises. Subjects will be advised to discontinue automated closed-loop insulin delivery and follow their usual insulin pump therapy for certain activities such as periods of strenuous exercise during the 7 day (phase 1) and 21 day (phase 2) home study phase.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM (conservatively adjusted for potential over-estimation). Secondary outcomes are the time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics. Safety evaluation comprises the tabulation of severe hypoglycaemic episodes.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 10 and 18 years of age (inclusive)
* The subject has type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative
* The subject/carer will have been an insulin pump user for at least 3 months, with good knowledge of insulin self-adjustment as judged by the investigator
* The subject/carer is willing to perform regular finger-prick blood glucose monitoring, with at least 4 blood glucose measurements taken every day
* HbA1c between 7.0% and 11.0 % (53 to 97mmol/mol) based on analysis from central laboratory or equivalent
* The subject is literate in English
* The subject is willing to wear closed-loop system at home and at school / college / work
* The subject is willing to follow study specific instructions

Exclusion Criteria:

* Non-type 1 diabetes mellitus including those secondary to chronic disease
* Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator.
* Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator
* Known or suspected allergy against insulin
* Subjects with clinically significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator
* Significantly reduced hypoglycaemia awareness as judged by the investigator
* Total daily insulin dose ≥ 2 IU/kg/day
* Total daily insulin dose <10 IU/day
* Reduced hypoglycaemia awareness
* Pregnancy, planned pregnancy or breast feeding
* Severe visual impairment
* Severe hearing impairment
* Subjects using implanted internal pacemaker
* Lack of reliable telephone facility for contact

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
The proportion of time spent in the target glucose range from 3.9 to 10.0 mmol/l based on CGM | 7 day (phase 1) and 21 day (phase 2) home study periods

SECONDARY OUTCOMES:
The proportion of time spent above and below the target glucose (3.9 to 10.0 mmol/l) based on CGM. | 7 day (phase 1) and 21 day (phase 2) home study periods
The proportion of time with glucose levels < 3.5 mmol/l and <2.8 mmol/l based on CGM | 7 day (phase 1) and 21 day (phase 2) home study periods
The proportion of time with glucose levels in significant hyperglycaemia, as based on CGM (glucose levels > 16.7 mmol/l) | 7 day (phase 1) and 21 day (phase 2) home study periods

OTHER OUTCOMES:
Safety evaluation | 7 day (phase 1) and 21 day (phase 2) home study periods
  Safety evaluation will comprise the number of episodes of hypoglycaemia, severe hypoglycaemia as well as nature and severity of any other adverse events, including ketone-positive hyperglycaemia.
Utility evaluation | 7 day (phase 1) and 21 day (phase 2) home study periods
  Utility of the system will be evaluated by the frequency and duration of use of the closed-loop system at home.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Director — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

REFERENCES:
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357
- [Background] Hovorka R, Kumareswaran K, Harris J, Allen JM, Elleri D, Xing D, Kollman C, Nodale M, Murphy HR, Dunger DB, Amiel SA, Heller SR, Wilinska ME, Evans ML. Overnight closed loop insulin delivery (artificial pancreas) in adults with type 1 diabetes: crossover randomised controlled studies. BMJ. 2011 Apr 13;342:d1855. doi: 10.1136/bmj.d1855. PMID 21493665
- [Background] Elleri D, Allen JM, Biagioni M, Kumareswaran K, Leelarathna L, Caldwell K, Nodale M, Wilinska ME, Acerini CL, Dunger DB, Hovorka R. Evaluation of a portable ambulatory prototype for automated overnight closed-loop insulin delivery in young people with type 1 diabetes. Pediatr Diabetes. 2012 Sep;13(6):449-53. doi: 10.1111/j.1399-5448.2012.00903.x. Epub 2012 Jul 23. PMID 22817340
- [Background] Kumareswaran K, Elleri D, Allen JM, Harris J, Xing D, Kollman C, Nodale M, Murphy HR, Amiel SA, Heller SR, Wilinska ME, Acerini CL, Evans ML, Dunger DB, Hovorka R. Meta-analysis of overnight closed-loop randomized studies in children and adults with type 1 diabetes: the Cambridge cohort. J Diabetes Sci Technol. 2011 Nov 1;5(6):1352-62. doi: 10.1177/193229681100500606. PMID 22226252
- [Result] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Stewart Z, Cheng P, Kollman C, Acerini CL, Dunger DB, Hovorka R. Day-and-Night Hybrid Closed-Loop Insulin Delivery in Adolescents With Type 1 Diabetes: A Free-Living, Randomized Clinical Trial. Diabetes Care. 2016 Jul;39(7):1168-74. doi: 10.2337/dc15-2078. Epub 2016 Jan 6. PMID 26740634
- [Result] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Acerini CL, Dunger DB, Hovorka R. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Suboptimally Controlled Adolescents With Type 1 Diabetes: A 3-Week, Free-Living, Randomized Crossover Trial. Diabetes Care. 2016 Nov;39(11):2019-2025. doi: 10.2337/dc16-1094. Epub 2016 Sep 9. PMID 27612500